CLINICAL TRIAL: NCT00210314
Title: Randomized Phase II Trial on Primary Chemotherapy With High-dose Methotrexate, Alone or Associated With High-dose Cytarabine, Followed by Response- and Age-tailored Radiotherapy for Immunocompetent Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: Phase II Trial of Combined Modality Treatment in Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: International Extranodal Lymphoma Study Group (IELSG), IELSG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG20
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Methotrexate; Cytarabine; Radiotherapy

ARMS (2):
- High-dose methotrexate alone (Active Comparator)
  Interventions: Drug: high dose methotrexate; Radiation: radiotherapy
- High-dose methotrexate associated with high dose cytarabine (Experimental)
  Interventions: Drug: high dose methotrexate; Drug: high dose cytarabine; Radiation: radiotherapy

INTERVENTIONS:
Drug: high dose methotrexate
Drug: high dose cytarabine
  Arms: High-dose methotrexate associated with high dose cytarabine
Radiation: radiotherapy

SUMMARY:
Aim of the study is to establish in a prospective, randomized clinical trial the activity of primary chemotherapy containing high dose-methotrexate, alone or combined with high dose cytarabine, in patients with primary central nervous system lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of non-Hodgkin's lymphoma.
2. Diagnostic sample obtained by stereotactic or surgical biopsy, CSF cytology examination or vitrectomy.
3. Disease exclusively localized into the central nervous system, cranial nerves or eyes.
4. Untreated patients (patients treated with steroids alone are eligible).
5. At least one measurable lesion.
6. Age 18 - 75 years.
7. ECOG performance status < 3
8. HBsAg-negative and Ab anti-HCV-negative serologic status.
9. No known HIV disease or immunodeficiency.
10. Adequate bone marrow (PLT > 100000 mm3, Hb ≥ 9 g/dl, ANC ≥ 2.000 mm3), renal (creatinine clearance ≥ 60 mL/min), cardiac (VEF ≥ 50%), and hepatic function (total serum bilirubin < 3 mg/dL, AST/ALT and gGT < 2 per upper normal limit value).
11. No previous or concurrent malignancies with the exception of surgically cured cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer and of other cancers without evidence of disease since at least 5 years (patients with a previous lymphoma diagnosis will be excluded).
12. Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
13. Non-pregnant and non-lactating status for female patients. Adequate contraceptive measures during study participation for sexually active patients of childbearing potential.
14. No concurrent treatment with other experimental drugs.
15. Informed consent signed by the patient before registration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-07; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The main endpoint is the complete remission (CR) rate after chemotherapy

SECONDARY OUTCOMES:
Overall response rate
Response duration (time to relapse or progression) for responder patients
Overall survival
Event-free survival
Meningeal relapse rate
Early and late neurotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Andres JM Ferreri, MD, Study Chair — Radiochemotherapy. San Raffaele Hospital. Milan; Michele Reni, MD, Study Chair — Radiochemotherapy. San Raffaele Hospital. Milan; Emanuele Zucca, MD, Study Chair — International Extranodal Lymphoma Study Group/Oncology Institute of Southern Switzerland (IOSI)
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland

REFERENCES:
- [Derived] Ferreri AJ, Reni M, Foppoli M, Martelli M, Pangalis GA, Frezzato M, Cabras MG, Fabbri A, Corazzelli G, Ilariucci F, Rossi G, Soffietti R, Stelitano C, Vallisa D, Zaja F, Zoppegno L, Aondio GM, Avvisati G, Balzarotti M, Brandes AA, Fajardo J, Gomez H, Guarini A, Pinotti G, Rigacci L, Uhlmann C, Picozzi P, Vezzulli P, Ponzoni M, Zucca E, Caligaris-Cappio F, Cavalli F; International Extranodal Lymphoma Study Group (IELSG). High-dose cytarabine plus high-dose methotrexate versus high-dose methotrexate alone in patients with primary CNS lymphoma: a randomised phase 2 trial. Lancet. 2009 Oct 31;374(9700):1512-20. doi: 10.1016/S0140-6736(09)61416-1. Epub 2009 Sep 18. PMID 19767089
- See also: Click here for more information about this study — http://www.ielsg.org